CLINICAL TRIAL: NCT01290133
Title: A Phase I, Randomized, Placebo-Controlled, Parallel-Group, Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Dose of the Captisol™ Formulation of Vestipitant (GW597599) in Healthy Adult Subjects
Brief Title: Single Dose Safety Study for Compound to Treat Post-Operative Nausea and Vomiting (PONV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Accenture (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VNK114995
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Post-Operative Nausea and Vomiting (PONV)
MeSH Terms: conditions — Vomiting | interventions — vestipitant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Drug (Experimental)
  Interventions: Drug: GW597599
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW597599 — Single dose IV infusion
  Arms: Active Drug
Drug: Placebo — Single dose IV infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to describe the safety and tolerability and pharmacokinetics of a single intravenous administration of the new, Sulfobutyl Ether-7-Beta-Cyclodextrin (Captisol™) based, formulation in Healthy Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
3. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 week will elapse between the cessation of HRT and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until after the follow-up visit and completion of all follow-up assessments or at least 7 days after study drug administration, whichever is longer.
4. Body weight greater than or equal to 50 kg and BMI less than or equal to 31 kg/m2.
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
6. QTcB or QTcF < 450 msec; or QTcB or QTcF < 480 msec in subjects with Bundle Branch Block.
7. AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

1. The subject has a positive pre-study drug screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
2. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
3. A positive test for HIV antibody.
4. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
5. History of regular alcohol consumption within 6 months of the study defined as:

   * an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
6. Smoking or regular use of tobacco- or nicotine-containing products within 2 weeks prior to screening.
7. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
8. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
9. History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinic uses heparin to maintain intravenous cannula patency).
10. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
11. Lactating females.
12. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
13. Unwillingness or inability to follow the procedures outlined in the protocol.
14. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
15. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
16. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
17. Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, Melbourne, Victoria, Australia